CLINICAL TRIAL: NCT03354013
Title: Genetic Screening and Investigating the Effect of Assisted Oocyte Activation in Couples with Diminished/aberrant Embryonic Development.
Brief Title: Genetic Screening and Assisted Oocyte Activation in Couples with Diminished/aberrant Embryonic Development.
Acronym: AOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B670201732853; 2017/0819 (Other: Commissie Medische Ethiek (UZ Gent))
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Embryo; Embryo Disorder; Genetic Disease
Keywords: AOA; embryo developmental problems; genetic screening; calcium pattern analysis
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AOA, genetic screening, calcium pattern (Experimental): Clinical setting: Patients will undergo ICSI-AOA. Furthermore, patients will give a saliva sample to do genetic screening. Genes important during oocyte activation and embryo development will be investigated.
  Also, calcium pattern analysis of the patients' spermatozoa will be executed.
  Interventions: Procedure: AOA; Diagnostic Test: Genetic screening; Diagnostic Test: Calcium pattern analysis

INTERVENTIONS:
Procedure: AOA — 100% ICSI-AOA will be performed.
Diagnostic Test: Genetic screening — Patients will donate a saliva sample. Genetic screening will take place for PLCzeta (male) and Dux4 (male and female). Also other possible genes involved in embryo development could be tested.
Diagnostic Test: Calcium pattern analysis — Male patients will donate a sperm sample. Calcium pattern analysis will take place by injecting the patients' sperm into mouse and/or human (in vitro matured) oocytes (research-donated control oocytes). This will estimate the sperm capability to induce calcium oscillations in the oocyte.

SUMMARY:
This is an interventional comparative study at the Department of Reproductive Medicine at Ghent University Hospital. Patients with previous embryo developmental problems are eligible for the study. Patients will undergo an ICSI-AOA treatment and will also be screened for genes important in the oocyte activation and embryonic development process. Also, the calcium releasing pattern of the patients' spermatozoa will be investigated.

DETAILED DESCRIPTION:
Assisted Oocyte Activation (ICSI-AOA) will be the treatment for these patients to overcome their previous embryo developmental problems. This protocol artificially induces calcium rises in the oocyte, which mimics the natural oocyte activation process induced by the sperm factor PLCzeta. If 6 or more mature oocytes are collected at oocyte retrieval, 50%ICSI and 50% ICSI-AOA will be applied to all oocytes. The best embryo(s) will be transferred back. Rest embryo(s) will be vitrified for future cycles. Patients will be followed up.

Furthermore, an additional sperm sample will be produced to investigate the calcium inducing pattern of the patients' spermatozoa. Thereby, mouse and/or human (research-donated control oocytes) will be pre-incubated with a Ca2+ sensitive dye. Next, human spermatozoa will be injected into these mouse/human oocytes and the calcium pattern will be recorded under an inverted epifluorescence microscope.

Both partners will give a saliva sample to screen for mutations possible genes involved in oocyte activation and embryo development.

ELIGIBILITY:
Inclusion Criteria:

* patients with one or more previous ICSI cycles (UZ Gent) AND
* patients with:
* complete developmental arrest (no transfer), or
* complete developmental delay (no morula/blastocyst on Day 5), or
* significantly reduced blastocyst formation (≤15%)
* willing and able to give informed consent

Exclusion Criteria:

* patients which went for oocyte or sperm donation
* patients with severe male infertility or low fertilization (<33%) after ICSI
* cycles requiring surgical sperm recovery procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Blastocyst rate | 5 days after oocyte retrieval
  Blastocyst rate will be calculated and blastocyst will be scored. The best quality embryos will be transferred and/or frozen.

SECONDARY OUTCOMES:
Pregnancy rate | Positive hCG 16 days after oocyte retrieval
  The level of beta-hCG in serum will be checked 16 days after oocyte retrieval
Live birth rate | 37 - 42 weeks after last menstruation
  Pregnant women will be followed up. Live births will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Petra De Sutter, M.D; PhD, Principal Investigator — University Ghent; Björn Heindryckx, Prof.; PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, East-Flandres, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cardona Barberan A, Bonte D, Boel A, Thys V, Paredis R, Machtelinckx F, De Sutter P, De Croo I, Leybaert L, Stoop D, Coucke P, Vanden Meerschaut F, Heindryckx B. Assisted oocyte activation does not overcome recurrent embryo developmental problems. Hum Reprod. 2023 May 2;38(5):872-885. doi: 10.1093/humrep/dead051. PMID 36931261